CLINICAL TRIAL: NCT01369810
Title: Outcome Study Following Reimbursement Changes in the Use of Fixed Combination Inhalers in Patients With Asthma or COPD in Iceland
Brief Title: Outcome Study Following Reimbursement Changes in the Use of Fixed Combination Inhalers in Patients With Asthma or Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RSE-DUM-2010/2
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
Keywords: Epidemiological; asthma; COPD; reimbursement; switch; outcomes associated with the change in reimbursement
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All patients who was on treatment with fixed combination asthma or COPD therapy by January 1 2010

SUMMARY:
To investigate how a switch from fixed combination treatment (ICS and LABA) to other treatments influence asthma or COPD treatment failure

ELIGIBILITY:
Inclusion Criteria:

* All patients who was on treatment with fixed combination asthma or COPD therapy by January 1 2010

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who was on treatment with fixed combination asthma or COPD therapy by January 1 2010
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2011-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To investigate how a switch from fixed combination treatment (ICS and LABA) to other treatments influence asthma or COPD treatment failure | Data will be extracted from the medical records and registries on one occassion, covering a period of 3 years

SECONDARY OUTCOMES:
To map out the development of asthma and COPD treatment in Iceland after the change in reimbursement | Data will be extracted from the medical records and registries on one occassion, covering a period of 3 years
To investigate health economic outcomes | Data will be extracted from the medical records and registries on one occassion, covering a period of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Unnur Steina Björnsdottir, MD, Principal Investigator — University of Iceland; Sveinbjörn Gizurason, Principal Investigator — University of Iceland; Georgios Stratelis, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Uppsala, Sweden